CLINICAL TRIAL: NCT00816829
Title: A 1-month, Randomized, Double-blind, Placebo-controlled Study of Fenofibrate 145 mg Tablet in Patients With Sleep Apnea Syndrome
Brief Title: Effect of Fenofibrate on Sleep Apnea Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was prematurely terminated because of slow recruitment
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Jean-Claude Ansquer, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C LF178P 05 01; 2005-000548-98
Record Dates: First submitted 2009-01-02; First posted 2009-01-05 (Estimated); Results first posted 2009-07-07 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2009-07

CONDITIONS: Dyslipidemia; Sleep Apnea Syndrome; Overweight; Obesity
Keywords: Dyslipidemia; Sleep Apnea Syndromes; Fenofibrate; Obese; Overweight or obese patients
MeSH Terms: conditions — Dyslipidemias; Sleep Apnea Syndromes; Overweight; Obesity | interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Fenofibrate-matching placebo tablet
  Interventions: Drug: Placebo
- 2 (Experimental): 145 mg NanoCrystal fenofibrate tablet
  Interventions: Drug: Fenofibrate

INTERVENTIONS:
Drug: Placebo — Fenofibrate-matching placebo tablet
  Arms: 1
Drug: Fenofibrate — 145 mg NanoCrystal tablet
  Arms: 2

SUMMARY:
Objectives: to investigate for the potential effect of fenofibrate on symptoms and biological changes associated with sleep apnea syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Having previous diagnosis of sleep apnea not treated with Continuous Positive Airway Pressure (CPAP) or presenting clinical symptoms of sleep apnea
* Overweight or obese, with BMI >= 25 kg/m² and < 40 kg/m².
* Known moderate hypertriglyceridemia, with fasting Triglycerides level >= 2.0 and < 6.0 mmol/L within 3 months before the inclusion.

Exclusion Criteria:

* indication for immediate CPAP
* other known endocrine disease, except treated and adequately controlled hypothyroidism
* renal failure or plasma creatinine level >130 µmol/L
* current chronic liver disease or ALanine Amino Transferase (ALT)> 2 times the upper normal limit (UNL)
* symptomatic gallbladder disease
* known muscular disease or creatine phosphokinase (CK) > 3 times UNL.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (1):
- Site 1, Paris, France

REFERENCES:
- [Derived] Bruckert E, Duchene E, Bonnefont-Rousselot D, Hansel B, Ansquer JC, Dubois A, Gaymard B. Proof of concept study: does fenofibrate have a role in sleep apnoea syndrome? Curr Med Res Opin. 2010 May;26(5):1185-92. doi: 10.1185/03007991003693581. PMID 20297950

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited and treated in a hospital in Paris between September 2005 and January 2008
Pre-assignment Details: In total 34 subjects were randomly allocated to treatment (i.e. Subjects Started). All the subjects received the study drug and completed the study. The study was prematurely terminated because of low recruitment.
Groups:
- Placebo: Placebo
- Fenofibrate: Fenofibrate 145 mg
Period: Overall Study
Arm/Group | Placebo | Fenofibrate
Started | 16 | 18
Completed | 16 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fenofibrate | Total
Number analyzed (Participants) | 16 | 18 | 34
Age Continuous [Mean (Standard Deviation); unit: years] | 55.2 (6.5) | 55.9 (5.4) | 55.6 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  France | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Obstructive Apneas
Description: Total number of obstructive apneas during sleep during one night after one month of treatment (i.e. an occlusion of the airways accompanied by ineffective respiratory efforts).
Time Frame: at one month of treatment
Population: The analysis was performed using the total sample of randomized subjects (16 on placebo and 18 on fenofibrate).
Measure: Median (Full Range); unit: Number of obstructive apneas
Arm/Group | Placebo | Fenofibrate
Number analyzed (Participants) | 16 | 18
Number of obstructive apneas | 30.5 [0 to 318] | 15.0 [0 to 168]
Statistical Analysis 1: Comparison: Placebo vs Fenofibrate; Comparison between groups was performed using an ANCOVA on log-transformed data at one month after the start of the treatment; Test type: Superiority or Other; p = 0.048, ANCOVA

2. Primary Outcome: Desaturations
Description: Total number of desaturation events (i.e. defined as a decrease by 3 - 4% in oxygen saturation) during sleep during one night after one month of treatment.
Time Frame: at one month of treatment
Population: The analysis was performed on the total sample of randomized subjects (16 on placebo and 18 in fenofibrate).
Measure: Median (Full Range); unit: Number of desaturations
Arm/Group | Placebo | Fenofibrate
Number analyzed (Participants) | 16 | 18
Number of desaturations | 171.0 [61.0 to 674.0] | 130.0 [14.0 to 219.0]
Statistical Analysis 1: Comparison: Placebo vs Fenofibrate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.203, ANCOVA

3. Primary Outcome: Sleep Time With Oxygen Saturation Below 90%
Description: Percentage of Sleep time with oxygen saturation below 90% (measured by oximetry). Marker of consequences of apneas/hypopneas on arterial oxygenation during sleep during one night after one month of treatment. Higher percentage are worst for the patients.
Time Frame: at one month of treatment
Population: The analysis was performed on the total sample of randomized subjects (16 on placebo and 18 on fenofibrate).
Measure: Median (Full Range); unit: Percentage of sleep time
Arm/Group | Placebo | Fenofibrate
Number analyzed (Participants) | 16 | 18
Percentage of sleep time | 11.5 [3.0 to 60.0] | 3.5 [0.0 to 49.0]
Statistical Analysis 1: Comparison: Placebo vs Fenofibrate; Comparison between groups was performed using Wilcoxon Test on data at one month after the start of the treatment; Test type: Superiority or Other; p = 0.007, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Apneas
Description: Total number of episodes of apneas (i.e. cessation of breathing for at least 10 seconds) from central, obstructive or mixed origin during sleep during one night after one month of treatment
Time Frame: at one month of treatment
Population: The analysis was performed on the total sample of randomized subjects (16 on placebo and 18 on fenofibrate).
Measure: Median (Full Range); unit: Number of apneas
Arm/Group | Placebo | Fenofibrate
Number analyzed (Participants) | 16 | 18
Number of apneas | 31.0 [0 to 617] | 20.5 [0 to 268]
Statistical Analysis 1: Comparison: Placebo vs Fenofibrate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.199, ANCOVA

5. Primary Outcome: Hypopneas
Description: Total number of episodes of hypopneas (i.e. 50% to 80% reduction in airflow with a decrease of 3-4% in arterial oxygen saturation) during sleep during one night after one month of treatment.
Time Frame: at one month of treatment
Population: The analysis was performed on the total sample of randomized subjects (16 on placebo and 18 on fenofibrate).
Measure: Median (Full Range); unit: Number of hypopneas
Arm/Group | Placebo | Fenofibrate
Number analyzed (Participants) | 16 | 18
Number of hypopneas | 69.5 [32.0 to 222.0] | 63.0 [1.0 to 179.0]
Statistical Analysis 1: Comparison: Placebo vs Fenofibrate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.114, ANCOVA

6. Primary Outcome: Index Apnea/Hypopnea
Description: Average number of apneas and/or hypopneas per hour of sleep during one night after one month of treatment.
Time Frame: at one month of treatment
Population: The analysis was performed on the total sample of randomized subjects (16 on placebo and 18 on fenofibrate).
Measure: Median (Full Range); unit: Number per hour of sleep
Arm/Group | Placebo | Fenofibrate
Number analyzed (Participants) | 16 | 18
Number per hour of sleep | 22.5 [4.0 to 114.0] | 17.0 [0 to 47.0]
Statistical Analysis 1: Comparison: Placebo vs Fenofibrate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.533, ANCOVA

7. Primary Outcome: Mixed Apneas
Description: Total number of mixed apneas (i.e. sleep apneas that have both obstructive and central component) during sleep during one night after one month of treatment.
Time Frame: at one month of treatment
Population: The analysis was performed on the total sample of randomized subjects (16 on placebo and 18 on fenofibrate).
Measure: Median (Full Range); unit: Number of mixed apneas
Arm/Group | Placebo | Fenofibrate
Number analyzed (Participants) | 16 | 18
Number of mixed apneas | 0.0 [0.0 to 220.0] | 1.0 [0.0 to 28.0]
Statistical Analysis 1: Comparison: Placebo vs Fenofibrate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.521, ANCOVA

8. Primary Outcome: Central Apneas
Description: Total number of central apneas (i.e. apneas with no respiratory effort present) during sleep during one night after one month of treatment.
Time Frame: at one month of treatment
Population: The analysis was performed on the total sample of randomized subjects (16 on placebo and 18 on fenofibrate).
Measure: Median (Full Range); unit: Number of central apneas
Arm/Group | Placebo | Fenofibrate
Number analyzed (Participants) | 16 | 18
Number of central apneas | 0.0 [0.0 to 68.0] | 1.0 [0.0 to 46.0]
Statistical Analysis 1: Comparison: Placebo vs Fenofibrate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.333, ANCOVA

9. Primary Outcome: Index of Apneas
Description: Average number of apneas per hour of sleep during one night after one month of treatment.
Time Frame: at one month of treatment
Population: The analysis was performed on the total sample of randomized subjects (16 on placebo and 18 on fenofibrate).
Measure: Median (Full Range); unit: Number per hour of sleep
Arm/Group | Placebo | Fenofibrate
Number analyzed (Participants) | 16 | 18
Number per hour of sleep | 4.0 [0.0 to 105.0] | 2.5 [0.0 to 45.0]
Statistical Analysis 1: Comparison: Placebo vs Fenofibrate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.264, ANCOVA

10. Primary Outcome: Index of Hypopneas
Description: Average number of hypopneas per hour of sleep during one night after one month of treatment.
Time Frame: at one month of treatment
Population: The analysis was performed on the total sample of randomized subjects (16 on placebo and 18 on fenofibrate).
Measure: Median (Full Range); unit: Number per hour of sleep
Arm/Group | Placebo | Fenofibrate
Number analyzed (Participants) | 16 | 18
Number per hour of sleep | 11.0 [4.0 to 31.0] | 9.5 [0.0 to 33.0]
Statistical Analysis 1: Comparison: Placebo vs Fenofibrate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.401, ANCOVA

ADVERSE EVENTS:
Arm/Group | Placebo | Fenofibrate
Serious Adverse Events (participants affected / at risk) | 0 | 1
Other Adverse Events (participants affected / at risk) | 1 | 3
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Placebo | Fenofibrate
Metabolic and medical procedures (Surgical and medical procedures) | 0/16 | 1/18
OTHER ADVERSE EVENTS (reported when occurring in more than 6.6% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Placebo | Fenofibrate
Back Pain (Musculoskeletal and connective tissue disorders) | 1/16 | 0/18
Cystitis (Infections and infestations) | 0/16 | 1/18
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 0/16 | 1/18
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0/16 | 1/18
Rash (Skin and subcutaneous tissue disorders) | 0/16 | 1/18
Abdominal distension (Gastrointestinal disorders) | 0/16 | 1/18

LIMITATIONS AND CAVEATS:
Only treatment emergent events have been presented. They are defined as events started at or after the 1st administration of study medication and includes events started prior to the 1st administration but which worsened after the 1st intake.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review.